CLINICAL TRIAL: NCT04826861
Title: Development and Implementation of Supporting Lifestyle Change in Obese Pregnant Mothers Through Wearable Internet-of-Things (SLIM) Intervention
Brief Title: Supporting Lifestyle Change in Obese Pregnant Mothers Through Wearable Internet-of-Things (SLIM)
Acronym: SLIM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Turku (Other)
Collaborators: University of California, Irvine (Other); Helsinki University Central Hospital (Other)
Responsible Party: Principal Investigator, Hannakaisa Niela-Vilen, PhD, Docent, University of Turku
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: SLIM
Record Dates: First submitted 2021-03-17; First posted 2021-04-01 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Pregnancy-Related Condition, Unspecified; Overweight or Obesity
Keywords: Pregnancy; Overweight; Obesity; Wearable Electronic Devices; Technology; Internet-Based Intervention
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention for overweight pregnant women (Other): Intervention will be delivered during antenatal visits in maternity care
  Interventions: Behavioral: SLIM intervention

INTERVENTIONS:
Behavioral: SLIM intervention — Core components: 1) goal setting, 2) motivational interviewing, 3) feedback, 4) health technology

SUMMARY:
Maternal obesity increases risks for the mother and her child. It is crucial to arouse the pregnant and postpartum women´s willingness of change and motivation to take care of their own and their unborn child´s health. Wearable devices can be helpful for weight-management, e.g. in improving participant's self-efficacy in making healthy behavior changes, improving self-awareness, in goal setting and getting feedback. More comprehensive research is required to implement the optimal weight-management intervention for overweight women during pregnancy and the postpartum period and to develop appropriate and feasible implementation strategies to support nurses to deliver interventions in maternity clinics.

The aim of this study is to evaluate the effectiveness of the Supporting Lifestyle Change in Obese Pregnant Mothers Through Wearable Internet-of-Things (SLIM) intervention. Secondary aim is to evaluate the implementation of SLIM intervention in maternity care.

Intervention was developed based on findings of overweight women and their care givers interview study. The intervention targeting overweight pregnant women to improve their weight-management will be delivered during routine perinatal visits from the first visit to three months after child birth. Interventions core components will be goalsetting, motivational interviewing, feedback and health technology. Health technology includes Oura-ring and ZotCare -application. ZotCare -application combines data from Oura Smart Ring, electronic food diary and it´s also platform for researchers to send e.g. questionnaires and surveys to participants. Oura-smartring is an advanced technology ring that monitors e.g. heart rate, heart rate variability (HRV), steps, body temperature and sleep) and a smartphone application that includes data from Oura, and electronic food diary. Data collected with Oura -smartrings will be transmitted to cloud servers via a smartphone. The cloud will be responsible for storing the data and for performing the data preprocessing and analysis methods. Interventions primary outcome will be self-efficacy. Secondary outcomes will be womens weight, depression symptoms, quality of life, pregnancy anxiety, perceived stress, sence of coherence and acceptability, appropriateness and feasibility of Intervention.

Data will be collected via Oura smartring, electronic food diary and validated measures: Weight Efficacy Life-Style Questionnaire (WEL), Self-Efficacy for Physical Activity Scale (PASE), six-factor questionnaire (6-FQ), Three Factor Eating Questionnaire (TFEQ-R18), WHOQOL-BREF, Sense of coherence (SOC-13), Pregnancy anxiety (PRAQ-R2), Perceived stress and Edinburgh Postnatal Depression scale (EPDS). Intervention implementation will be evaluated with process evaluation. Data will be collected from public health nurses working in maternity clinics using focus group interviews and workshops.

DETAILED DESCRIPTION:
Maternal obesity increases risks for the mother and her child. It is crucial to arouse the pregnant and postpartum women´s willingness of change and motivation to take care of their own and their unborn child´s health. Researchers have suggested that reﬁning the pre-existing prenatal care models, possibly incorporating diet and physical activity into interventions, could be useful. Continuous monitoring can provide real-time information between scheduled appointments and thus may be helpful for targeting and tailoring pregnancy follow-up. Wearable devices can be helpful for weight-management, e.g. in improving participant's self-efficacy in making healthy behavior changes, improving self-awareness, in goal setting and getting feedback. However, it's very important to identify and tailor the intervention into individual motivations in order to facilitate technology adoption. Technological solutions designed for the pregnant women, can balance the gap between limited resources and growing demand of maternity care service. More comprehensive research is required to implement the optimal weight-management intervention for overweight women during pregnancy and the postpartum period and to develop appropriate and feasible implementation strategies to support nurses to deliver interventions in maternity clinics.

The aim of this study is to evaluate the effectiveness of the Supporting Lifestyle Change in Obese Pregnant Mothers Through Wearable Internet-of-Things (SLIM) intervention. Secondary aim is to evaluate the implementation of SLIM intervention in maternity care.

Intervention was developed based on findings of overweight women and their care givers interview study. In addition, intervention was planned in collaboration with public health nurses working in maternity clinics in workshops. The intervention targeting overweight pregnant women to improve their weight-management will be delivered during routine perinatal visits from the first visit to three months after child birth. Interventions core components will be goalsetting, motivational interviewing, feedback and health technology. Health technology includes Oura-ring and ZotCare -application. ZotCare -application combines data from Oura Smart Ring, electronic food diary and it´s also platform for researchers to send e.g. questionnaires and surveys to participants. Oura-smartring is an advanced technology ring that monitors e.g. heart rate, heart rate variability (HRV), steps, body temperature and sleep) and a smartphone application that includes data from Oura, and electronic food diary. Data collected with Oura -smartrings will be transmitted to cloud servers via a smartphone. The cloud will be responsible for storing the data and for performing the data preprocessing and analysis methods. Interventions primary outcome will be self-efficacy. Secondary outcomes will be womens weight, depression symptoms, quality of life and sence of coherence.

Data will be collected via Oura smartring, electronic food diary and validated measures: Weight Efficacy Life-Style Questionnaire (WEL), Self-Efficacy for Physical Activity Scale (PASE), six-factor questionnaire (6-FQ), Three Factor Eating Questionnaire (TFEQ-R18), WHOQOL-BREF, Sense of coherence (SOC-13), Pregnancy anxiety (PRAQ-R2), Perceived stress and Edinburgh Postnatal Depression scale (EPDS). Intervention implementation will be evaluated with process evaluation. Interventions acceptability, appropriateness and feasibility will be assessed with validated measures: Acceptability of Intervention Measure (AIM), Intervention Appropriateness Measure (IAM), and Feasibility of Intervention Measure (FIM). Data will be collected from public health nurses working in maternity clinics using focus group interviews and workshops.

ELIGIBILITY:
Inclusion Criteria:

* pregnancy maximum 15 gestational weeks
* BMI >25
* finnish language

Exclusion Criteria:

* women who don´t have smart device
* severe mental illness (such as schizophrenia)
* diabetes mellitus type 1
* limitation of motility

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 55 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2023-05-15 (Actual); Study Completion 2023-05-15 (Actual)

PRIMARY OUTCOMES:
Change of eating self-efficacy of overweight women | Change from first trimester Self-efficacy at third trimester and further at two months after delivery
  Validated measurement tool:
  Weight Efficacy Life-Style Questionnaire (WEL) The 20-item questionnaire asks participants to rate their confidence in their ability to avoid eating on a 10-point Likert scale, 0 (not confident) to 9 (very confident). Scores range from 0 to 180 with higher scores indicating greater levels of self-efficacy.
Change of physical activity self-efficacy of overweight women | Change from first trimester Self-efficacy at third trimester and further at two months after delivery
  Validated measurement tool:
  Self-Efficacy for Physical Activity Scale (PASE). The 5-item questionnaire asks participants to rate their confidence in their ability to regular physical activity on a 5-point Likert scale, 1 (not confident) to 5 (very confident). Scores range from 5 to 25 with higher scores indicating greater levels of self-efficacy.

SECONDARY OUTCOMES:
Weight during pregnancy and after delivery | Through study completion, an average of 11 to 12 months.
  Measurement: Womens weight (patient records)
Change of depression symptoms of overweight women | From first trimester depression symptoms at third trimester and further at two months after delivery
  Validated measurement tool:
  Perceived stress and Edinburgh Postnatal Depression scale (EPDS). The 10-item questionnaire asks participants to rate their depression symptoms on a 4-point Likert scale. Scores range from 0 to 30 with higher scores indicating greater levels of depression.
Change of overweight womens quality of life | Change from first trimester quality of life at third trimester and further at two months after delivery
  Validated measurement tool:
  WHO quality of life (WHOQOL-BREF). The 26-item questionnaire asks participants to rate their quality of life on a 5-point Likert scale, 1 to 5. Scores range from 0 to 100 with higher scores indicating better quality of life.
Change of overweight womens sense of coherence | Change from first trimester sence of coherence at third trimester and further at two months after delivery
  Validated measurement tool:
  Sense of coherence (SOC-13).
  The 13-item questionnaire asks participants to rate their sence of coherence on a 7-point Likert scale, 1 to 7. Higher scores indicate better sence of coherence.
Change of pregnancy anxiety. | Change from first trimester anxiety at third trimester and further at two months after delivery
  Validated tool:
  Pregnancy anxiety questionnaire-revised for all pregnant women regardless of parity:(PRAQ-R2) The 10-item questionnaire asks participants to rate their pregnancy anxiety on a 5-point Likert scale, 1 to 5. Higher scores indicate higher pregnancy anxiety.
Change of perceived stress | Change from first trimester perceived stress at third trimester and further at two months after delivery
  Validated tool: A global measure of perceived stress (original versions). The 10-item questionnaire asks participants to rate their pregnancy anxiety on a 5-point Likert scale, 1 to 5. Higher scores indicate higher perceived stress.
Interventions acceptability, appropriateness and feasibility | At gestational week 20, 34 and three months after delivery
  Validated measures: Acceptability of Intervention Measure (AIM), Intervention Appropriateness Measure (IAM) and Feasibility of Intervention Measure (FIM).
  The 15-item questionnaire asks participants to rate interventions acceptability, appropriateness and feasibility on a 5-point Likert scale, 1 to 5. Higher scores indicate higher acceptability, appropriateness and feasibility.

CONTACTS AND LOCATIONS:
Overall Officials: Hannakaisa Niela-vilen, PhD, Principal Investigator — University of Turku
Locations (1):
- Maternity care unit, Loimaa, Finland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Saarikko J, Axelin A, Huvinen E, Rahmani AM, Kolari T, Niela-Vilen H. Effectiveness of supporting lifestyle change in pregnant mothers with obesity through the wearable internet-of-things (SLIM) -intervention on self-efficacy in weight management in pregnant women: A quasi-experimental trial. Midwifery. 2025 Jan;140:104235. doi: 10.1016/j.midw.2024.104235. Epub 2024 Nov 9. PMID 39549539
- [Derived] Saarikko J, Axelin A, Huvinen E, Rahmani AM, Azimi I, Pasanen M, Niela-Vilen H. Supporting lifestyle change in obese pregnant mothers through the wearable internet-of-things (SLIM) -intervention for overweight pregnant women: Study protocol for a quasi-experimental trial. PLoS One. 2023 Jan 19;18(1):e0279696. doi: 10.1371/journal.pone.0279696. eCollection 2023. PMID 36656819